CLINICAL TRIAL: NCT05599399
Title: Impact of Gum Acacia on Gut-microbiota Derived Metabolites in Chronic Kidney Disease Patients
Brief Title: Impact of Gum Acacia on Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0107213
Record Dates: First submitted 2022-10-14; First posted 2022-10-31 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-09

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Gum Arabic

STUDY DESIGN:
Intervention Model Description: Open labelled, prospective, two-arm, parallel group, non-placebo controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients receiving gum acacia (Active Comparator): Group one will receive gum acacia extract as an add-on therapy on daily basis
  Interventions: Dietary Supplement: Gum acacia
- Patients receiving no intervention (No Intervention): Group two will not receive add-on therapy; they will receive standard care only.

INTERVENTIONS:
Dietary Supplement: Gum acacia — 25 grams of gum acacia powder is administered on daily-basis
  Arms: Patients receiving gum acacia

SUMMARY:
The aim of the study is to evaluate the impact of gum acacia on serum levels of protein-bound uremic toxins (indoxyl sulfate and p-cresyl sulfate).In addition to the evaluation of its effect on metabolic profile and disease progression in chronic kidney disease patients.

DETAILED DESCRIPTION:
1. Ethical committee approval has been obtained from Ethics committee of Faculty of Medicine, Alexandria University.
2. All participants should agree to take part in this clinical study and will provide informed consent.
3. Eighty chronic kidney disease patients,will be recruited from the Kidney and Urology Center (KUC) and Alexandria main university hospital (AMUH).

   The 80 participants will be randomly assigned into 2 arms.

   Control arm (n=40): will be treated with standard treatment without any herbal intervention.

   Intervention arm (n=40): will be treated with standard treatment in addition to gum acacia sachets. Each sachet contains 25 g of gum acacia powder to be taken on daily-basis for 3 months.
4. All patients will be submitted to :

   * Full patient history and clinical examination.
   * Blood withdrawal in order to conduct lab work.
5. Patients demographic data will be recorded with respect to age, weight and other co-morbidities.
6. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
7. Results, conclusion, discussion and recommendations will be given.

ELIGIBILITY:
Inclusion Criteria:

* Non-hemodialysis CKD patients (Stage III -V)
* Age: above 18 years

Exclusion Criteria:

* Hemodialysis patients
* Pregnancy & lactation
* Patients recently treated with antibiotic regimen (2 - 4 weeks)
* Malignancy
* Inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline values of renal profile of chronic kidney disease patients. | 3 months
  Suggested parameters include: urea, serum creatinine, uric acid, urinary Albumin to creatinine (ACR)
Percentage change from baseline scores of serum levels of suggested gut-derived protein bound uremic toxins | 3 months
  indoxyl sulfate, p-cresyl sulfate sulfate)
Mean change from baseline values of complete blood picture | 3 months
  Suggested parameters include: Haemoglobin (Hb) , White blood cells count (WCC), Platelets count (PLT)
Mean change from baseline values of serum electrolytes levels | 3 months
  Suggested parameters include: serum sodium, serum potassium, serum calcium and serum phosphorus
Mean change from baseline values of serum albumin levels | 3 months
  Suggested parameters include: serum albumin

SECONDARY OUTCOMES:
Effect of gum acacia on disease progression | 3 months
  expressed in terms of loss 50% in glomerular filtration rate and need for renal replacement therapy loss 50% in glomerular filtration rate and need for renal replacement therapy
Adverse effects of gum acacia will be also addressed through adverse effect monitoring system. monitoring system | 3 months
  Patients will be contacted on a regular basis to monitor adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Merna M. AbouKhatwa, BSc, Principal Investigator — Faculty of Pharmacy, Alexandria University
Locations (1):
- Kidney and Urology Center (KUC), Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No